CLINICAL TRIAL: NCT03903614
Title: Handwriting Intervention, With vs. Without a Rightward Bias, in a Junior High School-A Randomized Controlled Study
Brief Title: Sensory Motor Lateralization as Handwriting Intervention in School-Based OT
Acronym: SML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary H. Teng (Other)
Responsible Party: Sponsor-Investigator, Mary H. Teng, Principal Investigator, Teng, Mary H.
Organization: Teng, Mary H. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TengM; Conventional School-Based OT (Other: TengM); NCT03514992 (obsolete NCT alias)
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Developmental Dysgraphia
Keywords: Developmental Dysgraphia; Ambidexterity; Outcome study
MeSH Terms: conditions — Agraphia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, since the Principal Investigator was the intervener to both study groups, and also the data collector, an effort was made to ensure that both the pre- and posttest were administered in the presence of one other Occupational Therapist, Registered (OTR) and/or a Physical Therapist, who shared the use of the room with Mrs. Teng, test booklets were encrypted, and, that the participants, parents, test graders (one different OTR to each test instrument), and statisticians were kept blind to the group assignment of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory Motor Lateralization (SML) (Experimental): This was a group of 8 junior high school students who received SML in school for handwriting difficulty during the 2012-13 School Year. The participants received left eye-and-ear occlusion, fitness exercises, fine motor speed training, and handwriting practice on their right hand only.
  Interventions: Behavioral: SML
- Conventional School-Based OT (CON) (Active Comparator): This was a group of 8 junior high school students who received conventional school-based Occupational Therapy service for handwriting difficulty during the 2012-13 School Year. The participants received a like fitness exercises, fine motor speed training, and handwriting practice on their dominant hand instead.
  Interventions: Behavioral: CON

INTERVENTIONS:
Behavioral: SML — SML consists of supervised handwriting practice, fitness exercises, and fine motor speed drills that preferentially belabor a participant's right eye, ear, hand and leg during therapy.
  Other Names: Cerebral Lateralization Intervention
  Arms: Sensory Motor Lateralization (SML)
Behavioral: CON — CON consists of supervised handwriting practice, fitness exercises, and fine motor speed drills on the participant's dominant hand.
  Other Names: Conventional School-Based OT
  Arms: Conventional School-Based OT (CON)

SUMMARY:
Children who attend School-Based Occupational Therapy (SBOT) show mixed dominance and a liable decreased in the structural and functional differentiation between the two hemispheres. The lack of right-left disparity has been found to link to mirror invariance, poor spatial organization, fragmentary reversals, and handwriting difficulty. This study intends to find out, whether, Sensory Motor Lateralization (SML), "With" a rightward bias, profits handwriting more than the conventional (CON) "Without".

DETAILED DESCRIPTION:
10 to 30% of school children suffer handwriting difficulty. Many of them are eventually referred to SBOT for remedial intervention. Among these children, 70% show mixed dominance in their hand and/or leg use, and a likely functional and structural interhemispherical asymmetry reduction. This would make them right-left symmetrical. Learning, thus, may be challenged, because people who are right-left balanced would not have a consistent reference point to process the learning materials regularly in any pre-determined directions. They are, thus, prone to suffer mirror invariance, fragmentary reversal errors, and handwriting difficulty, especially with the fast and accurate construction of asymmetrical letters from memory.

To enhance right-left disparity, dispel mirror invariance, and facilitate the automatized handwriting, SML preferentially belabors one's right eye, ear, hand and leg in therapy, that would greater engage the left hemisphere for its acclaimed vantages over learning. This study investigates, whether SML, wielding such a rightward bias, profits handwriting greater than CON.

ELIGIBILITY:
Inclusion Criteria:

* Any Special or Regular Education students with Individualized Education Plans (IEPs), OT mandates, and handwriting goals.
* Has Intelligence Quotient (IQ) equal to or above 60.
* Ambulatory.
* Proficient in English, and fluent in naming, identifying, and accessing the sequence of letters in the alphabet.
* The students who attend Physical Therapy (PT), Adaptive Physical Education (PE), and any other programs are included, if the programs being provided are skill-, theme-, or task-oriented, not involving any muscle strengthening activities.

Exclusion Criteria:

* All are excluded, if the study candidates have any medical condition(s) that would prohibit them from the full physical participation in school.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2013-01-04 (Actual); Study Completion 2013-06-12 (Actual)

PRIMARY OUTCOMES:
SML excels CON in manuscript letter legibility | Change from Baseline percent accuracy score at 3 months
  Assess by the percent accuracy score of manuscript letter legibility derived from the Wold Sentence Copying Test (WSCT). TThe letter legibility score was calculated by counting the total number of letters the participant wrote minus the writing errors per THS-R criteria, divided by the total number of characters written, and multiplied by 100. The minimum is 0, and the maximum is 100. The higher values represent better treatment outcome.
SML excels CON in script letter legibility | Change from Baseline percent accuracy score at 3 months
  Assess by the percent accuracy score of script letter legibility derived from the Wold Sentence Copying Test (WSCT). The letter legibility score was calculated by counting the total number of letters the participant wrote minus the writing errors per THS-R criteria, divided by the total number of characters written, and multiplied by 100. The minimum is 0, and the maximum is 100. The higher values represent better treatment outcome.
SML excels CON in manuscript transcription speed | Change from Baseline letters per minute at 3 months
  Assess by WSCT.Speed was derived from the total number of letters written timed 60, divided by the total number of seconds used, and recorded as number of letters per minute. The minimum is 0, and there is no maximum. The higher values represent better treatment outcome.
SML excels CON in script transcription speed | Change from Baseline letters per minute at 3 months
  Assess by WSCT. Speed was derived from the total number of letters written timed 60, divided by the total number of seconds used, and recorded as number of letters per minute. The minimum is 0, and there is no maximum. The higher values represent better treatment outcome.

OTHER OUTCOMES:
SML excels CON in Visual Motor Integration | Change from Baseline raw score at 3 months
  Assess by the Developmental Test of Visual Motor Integration (DTVMI). The minimum is 0, and the highest is 30. The higher scores represent better treatment outcome
SML excels CON in Visual Perception | Change from Baseline raw score at 3 months
  Assess by the Developmental Test of Visual Motor Integration (DTVMI). The minimum is 0, and the highest is 30. The higher scores represent better treatment outcome.
SML excels CON in Motor Coordination | Change from Baseline raw score at 3 months
  Assess by the Developmental Test of Visual Motor Integration (DTVMI). The minimum is 0, and the highest is 30. The higher scores represent better treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mary H Teng, MS, OTR, Principal Investigator

IPD SHARING:
Plan to Share IPD: Yes
I intend to publish this study. I'll make individual participant data (IPD) available to other researchers afterwards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: I intend to publish this study. I'll make IPD available to other researchers afterwards.
Access Criteria: I intend to publish this study. I'll make IPD available to other researchers afterwards.

REFERENCES:
- [Background] Adi-Japha E, Landau YE, Frenkel L, Teicher M, Gross-Tsur V, Shalev RS. ADHD and dysgraphia: underlying mechanisms. Cortex. 2007 Aug;43(6):700-9. doi: 10.1016/s0010-9452(08)70499-4. PMID 17710822
- [Background] Anguera JA, Russell CA, Noll DC, Seidler RD. Neural correlates associated with intermanual transfer of sensorimotor adaptation. Brain Res. 2007 Dec 14;1185:136-51. doi: 10.1016/j.brainres.2007.09.088. Epub 2007 Oct 11. PMID 17996854
- [Background] Assmus A, Marshall JC, Noth J, Zilles K, Fink GR. Difficulty of perceptual spatiotemporal integration modulates the neural activity of left inferior parietal cortex. Neuroscience. 2005;132(4):923-7. doi: 10.1016/j.neuroscience.2005.01.047. PMID 15857698
- [Background] Bryden PJ, Bruyn J, Fletcher P. Handedness and health: an examination of the association between different handedness classifications and health disorders. Laterality. 2005 Sep;10(5):429-40. doi: 10.1080/13576500442000193. PMID 16191813
- [Background] Coghill RC, Gilron I, Iadarola MJ. Hemispheric lateralization of somatosensory processing. J Neurophysiol. 2001 Jun;85(6):2602-12. doi: 10.1152/jn.2001.85.6.2602. PMID 11387404
- [Background] Corbetta M, Shulman GL. Control of goal-directed and stimulus-driven attention in the brain. Nat Rev Neurosci. 2002 Mar;3(3):201-15. doi: 10.1038/nrn755. PMID 11994752
- [Background] Davidson RJ, Jackson DC, Kalin NH. Emotion, plasticity, context, and regulation: perspectives from affective neuroscience. Psychol Bull. 2000 Nov;126(6):890-909. doi: 10.1037/0033-2909.126.6.890. PMID 11107881
- [Background] Hirnstein M, Bayer U, Ellison A, Hausmann M. TMS over the left angular gyrus impairs the ability to discriminate left from right. Neuropsychologia. 2011 Jan;49(1):29-33. doi: 10.1016/j.neuropsychologia.2010.10.028. Epub 2010 Oct 28. PMID 21035475
- [Background] Hirnstein M, Hugdahl K, Hausmann M. How brain asymmetry relates to performance - a large-scale dichotic listening study. Front Psychol. 2014 Jan 2;4:997. doi: 10.3389/fpsyg.2013.00997. eCollection 2014. PMID 24427151
- [Background] Hoy MM, Egan MY, Feder KP. A systematic review of interventions to improve handwriting. Can J Occup Ther. 2011 Feb;78(1):13-25. doi: 10.2182/cjot.2011.78.1.3. PMID 21395194
- [Background] Hughes CM, Reissig P, Seegelke C. Motor planning and execution in left- and right-handed individuals during a bimanual grasping and placing task. Acta Psychol (Amst). 2011 Sep;138(1):111-8. doi: 10.1016/j.actpsy.2011.05.013. Epub 2011 Jun 12. PMID 21663882
- [Background] Dundas EM, Plaut DC, Behrmann M. The joint development of hemispheric lateralization for words and faces. J Exp Psychol Gen. 2013 May;142(2):348-58. doi: 10.1037/a0029503. Epub 2012 Aug 6. PMID 22866684
- [Background] Hlustik P, Solodkin A, Gullapalli RP, Noll DC, Small SL. Functional lateralization of the human premotor cortex during sequential movements. Brain Cogn. 2002 Jun;49(1):54-62. doi: 10.1006/brcg.2001.1483. PMID 12027392
- [Background] Jancke L. A differential effect of concurrent verbal activity on right arm movements rightwards and leftwards. Cortex. 1993 Mar;29(1):161-6. doi: 10.1016/s0010-9452(13)80221-3. PMID 8472554
- [Background] Granert O, Peller M, Gaser C, Groppa S, Hallett M, Knutzen A, Deuschl G, Zeuner KE, Siebner HR. Manual activity shapes structure and function in contralateral human motor hand area. Neuroimage. 2011 Jan 1;54(1):32-41. doi: 10.1016/j.neuroimage.2010.08.013. Epub 2010 Aug 12. PMID 20708692
- [Background] Schott GD. Mirror writing: neurological reflections on an unusual phenomenon. J Neurol Neurosurg Psychiatry. 2007 Jan;78(1):5-13. doi: 10.1136/jnnp.2006.094870. Epub 2006 Sep 8. PMID 16963501
- [Background] Sabate M, Gonzalez B, Rodriguez M. Brain lateralization of motor imagery: motor planning asymmetry as a cause of movement lateralization. Neuropsychologia. 2004;42(8):1041-9. doi: 10.1016/j.neuropsychologia.2003.12.015. PMID 15093143
- [Background] Saugstad LF. Cerebral lateralisation and rate of maturation. Int J Psychophysiol. 1998 Jan;28(1):37-62. doi: 10.1016/s0167-8760(97)00063-9. PMID 9506310
- [Background] Lee DR, Kim YH, Kim DA, Lee JA, Hwang PW, Lee MJ, You SH. Innovative strength training-induced neuroplasticity and increased muscle size and strength in children with spastic cerebral palsy: an experimenter-blind case study--three-month follow-up. NeuroRehabilitation. 2014;35(1):131-6. doi: 10.3233/NRE-131036. PMID 24419014
- [Background] Mazziotta JC, Phelps ME. Human sensory stimulation and deprivation: positron emission tomographic results and strategies. Ann Neurol. 1984;15 Suppl:S50-60. doi: 10.1002/ana.410150711. PMID 6611127
- [Background] Peters M, Reimers S, Manning JT. Hand preference for writing and associations with selected demographic and behavioral variables in 255,100 subjects: the BBC internet study. Brain Cogn. 2006 Nov;62(2):177-89. doi: 10.1016/j.bandc.2006.04.005. Epub 2006 Jun 23. PMID 16797814
- [Background] Vingerhoets G, Acke F, Alderweireldt AS, Nys J, Vandemaele P, Achten E. Cerebral lateralization of praxis in right- and left-handedness: same pattern, different strength. Hum Brain Mapp. 2012 Apr;33(4):763-77. doi: 10.1002/hbm.21247. Epub 2011 Apr 15. PMID 21500314
- [Background] Vingerhoets G, Sarrechia I. Individual differences in degree of handedness and somesthetic asymmetry predict individual differences in left-right confusion. Behav Brain Res. 2009 Dec 1;204(1):212-6. doi: 10.1016/j.bbr.2009.06.004. Epub 2009 Jun 10. PMID 19523492
- See also: Bédard, P., Wu, M., & Sanes, J. N. (2011). Brain Activation Related to Combinations of Gaze Position, Visual Input, and Goal-Directed Hand Movements. Cerebral Cortex, 21(6), 1273-1282. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3097986/
- See also: Corballis, M. C. (2014). Left brain, right brain: facts and fantasies. PLoS Biology, 12(1), e1001767. — https://doi.org/10.1371/journal.pbio.1001767
- See also: Frey, S. H. (2008). Tool use, communicative gesture and cerebral asymmetries in the modern human brain. Archives of Philosophical Transactions of the Royal Society of London Biological Sciences, 363, 1951-7. — http://rstb.royalsocietypublishing.org/content/royptb/363/1499/1951.full.pdf
- See also: Guerraz, M., Blouin, J., & Vercher, J. L. (2003). From head orientation to head control: evidence of both neck and vestibular involvement in hand drawing. Experimental Brain research, 150, 40-9. — https://link.springer.com/article/10.1007/s00221-003-1411-y
- See also: Heilman, K. M., Howell, G., Valenstein, E., & Rothi, L. (1980). Mirror-reading and writing in association with right-left spatial disorientation. Journal of Neurology, Neurosurgery, and Psychiatry, 43(9), 774-80. — http://dx.doi.org/10.1136/jnnp.43.9.774
- See also: Sibley, B. A. and Jennifer L. Etnier, J. L. (2003). The relationship between physical activity and cognition in children: A meta-analysis. Review Article. Pediatric Exercise Science, 15, 243-256. — https://journals.humankinetics.com/doi/abs/10.1123/pes.15.3.243
- See also: Weintraub, N., & Graham, S. (2000). The contribution of gender, orthographic, finger function, and visual-motor processes to the prediction of handwriting status. The Occupational Therapy Journal of Research, 20(2), 121-140 — http://journals.sagepub.com/doi/abs/10.1177/153944920002000203